CLINICAL TRIAL: NCT06666257
Title: Continuous Glucose and E-Monitoring to Support Healthy Weight Gain in Pregnancies - The GEM Study
Acronym: GEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lisa Jansen, Assistant Professor, Arkansas Children's Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 276728; 5P20GM109096 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pregnancies at Increased Risk for Excessive Gestational Weight Gain; Ecological Momentary Assessment and Intervention; Continuous Glucose Monitor
Keywords: Pregnancy; Obesity; Continuous Glucose Monitoring; Ecological Momentary Intervention; Gestational Weight Gain; Overweight
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Overweight | interventions — Pregnancy

STUDY DESIGN:
Intervention Model Description: This pilot study tests the feasibility of a single-arm, remotely delivered behavioral lifestyle intervention program for pregnant women with overweight and obesity. Modeled after the SmartMoms approach, the program combined weekly virtual health coach sessions with motivational interview techniques, daily weight and activity tracking, continuous glucose monitoring, and tailored education to support healthy gestational weight gain. A simulated control arm will be created from existing datasets for preliminary comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote Weight & Step Monitoring + CGM (Experimental): Women will engage in the remote intervention resembling efforts used by the SmartMoms intervention, but adapted to the needs of Arkansas women while also wearing unblinded CGM devices providing insights to glycemic trends in response to lifestyle factors.
  Interventions: Behavioral: Continuous Glucose and E-Monitoring to Support Healthy Weight Gain in Pregnancy

INTERVENTIONS:
Behavioral: Continuous Glucose and E-Monitoring to Support Healthy Weight Gain in Pregnancy — The intervention we are basing our adaptations on is a ecological momentary intervention, meaning it is integrated into participants daily lifestyle and schedule. Using an established framework for tracking daily body weight and physical activity, a gestational weight gain trajectory is estimated. Based on the data, recommendation prompts for exercise and diet will be discussed with participants during motivational interviewing. For the CGM piece, participants will wear unblinded CGM devices and have access to CGM linked app features that allow insights and reactivity to personal glycemic data

SUMMARY:
This single-arm pilot study will evaluate the feasibility and acceptability of a remotely delivered behavioral lifestyle intervention, adapted from the SmartMoms framework, to promote health gestational weight gain in pregnant women with overweight and obesity. Twelve to sixteen participants will receive weekly virtual motivational interview sessions with trained health coaches, review their daily weight data, step count, and continuous glucose monitoring data, and tailored guidance on physical activity and nutrition. Educational content will be delivered electronically, with peer support provided through a closed online group. A simulated (mock) control arm will be created post hoc from existing records for preliminary comparisons; all enrolled participants will receive the intervention.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility of delivering a remotely administered behavioral lifestyle intervention for pregnant women with overweight and obesity, adapted from the established SmartMoms framework, using a simulated (mock) control arm for comparison. This pilot study will enroll approximately 12-16 participants and will focus on evaluating feasibility, acceptability, and preliminary signals of impact to inform a future randomized controlled trial.

The intervention is tailored to the needs of women in Arkansas and aims to promote healthy gestational weight gain through motivational interviewing, physical activity promotion, education on dietary recommendations and self-monitoring. Participants will be encouraged to meet current pregnancy exercise guidelines (>= 30 minutes of moderate-intensity activity on most, if not all days) and to follow a balanced diet consistent with caloric intake recommendations for appropriate gestational weight gain based on individual pre-pregnancy BMI.

Each participant will be provided with an internet connected bodyweight scal, and pedometer for daily self-monitoring. These devices will automatically transmit weight and step data to the study team. Participants will also wear a continuous glucose monitor (CGM) throughout their pregnancy to track temporal glucose patterns, which will be reviewed with the study's registered dietitian (RD) and health coaches.

Intervention delivery will include weekly virtual motivational interview sessions with a trained health coach. Sessions will review weight gain trajectory, dietary intake, physical activity patterns, and CGM data, and will provide tailored behavioral strategies for meeting gestational weight gain goals. Educational materials will be delivered electronically to participants' smartphones. A closed online forum will be available for peer support, following the SmartMoms framework.

The simulated control arm will be generated post hoc by matching trial participants to publicly available datasets based on gestational age, BMI category, and other relevant covariates. This mock control will serve only as a comparator for preliminary analyses; all enrolled participants will receive the active intervention.

The intervention will begin between 16-20 weeks' gestation and continue until delivery (20-24 weeks per participant). All motivational interviewing sessions will be delivered remotely, and participants will be trained individually on safe and effective use of study tools.

ELIGIBILITY:
The formative phase (Phase I), classified as exempt by the institutional review board will seek participation from individuals meeting the following criteria:

1. Currently pregnant or pregnant within the past 36 months.
2. Community partners with relevant perspectives to inform recruitment, adaptation approaches and feasibility of the phase 2 pilot trial.

Clinical Trial (Phase 2)

Inclusion Criteria:

* pregnant women less than 20 weeks of gestation at time of screening
* 18-45 years of age
* BMI of 25 - 40 kg/m-2
* Expecting a singleton pregnancy
* Smartphone and/or reliable internet access
* Willing to be identifiable to other study participants in the study program .

Exclusion Criteria:

* Smoker
* Preexisting medical conditions that might be exacerbated by pregnancy (e.g., diabetes mellitus, chronic renal failure, hypertension, malignancies, seizure disorder, lupus, drug or alcohol abuse, serious psychiatric disorders)
* Current mental health or eating disorder
* Contraindication to exercise (OB/GYN release is obtained prior to consent)
* Conceived with assisted fertility treatments
* Medications during pregnancy known to influence fetal growth (e.g., thyroid hormone, glucocorticoids, insulin, oral hypoglycemic agents)
* Plans to move out of the state in the next 6 months following screening.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility data of the modified EMI: AR-GEM Study - Recruitment and Retention | continuous, from study enrollment at 16-20 weeks until study completion, an average of 6 months
  Maternal recruitment and retention rates (total number of participants recruited and retained)
Feasibility data of the modified EMI: SmartMomsAR - Acceptability | continuous, from study enrollment at 16-20 weeks until study completion, an average of 6 months
  Acceptability scores from online intervention satisfaction questionnaires, 5 point Likert Scale system
Feasibility data of the modified EMI: SmartMomsAR - Protocol Adherence | continuous, from study enrollment at 16-20 weeks until study completion, an average of 6 months
  Adherence to study protocol via process measures. (Percentage of complete data points)

SECONDARY OUTCOMES:
Incidence of appropriate gestational weight gain per 2009 NASM guidelines. | data is derived through study completion, an average of 6 months.
  Frequencies (percentage) of appropriate gestational weight gain incidence. Maternal weight (lbs) over time.
Change in healthful lifestyle behaviors - HEI | data is derived through study completion, an average of 6 months.
  Change scores for healthy eating index (HEI)
Change in healthful lifestyle behaviors - Steps (Physical Activity) | data is derived through study completion, an average of 6 months.
  Change scores for physical activity counts (steps) as assessed commercial accelerometer.
Change in healthful lifestyle behaviors - Glycemic profile | data is derived through study completion, an average of 6 months.
  Summary of glycemic profile data (mg/dL) as assessed by CGM.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa T Jansen, PhD, Principal Investigator — Arkansas Children's Hospital Research Institute; University of Arkansas for Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 21 days of having IRB approval for the finalized phase II protocol (anticipated to be available 05/01/25)
Access Criteria: Individual participant data (IPD) from this feasibility pilot study will be shared with qualified researchers conducting analyses that align with the study's objectives, specifically in relation to [study-specific areas of interest, e.g., behavior modification in pregnancy, glucose metabolism, etc.]. All data requests must include a detailed research proposal outlining planned analyses and the statistical methods. Proposals will be reviewed by the Principal Investigator and an independent review board for scientific validity, ethical considerations, and alignment with study objectives. A Data Sharing Agreement (DSA) must be signed prior to data release. Documents can be submitted via [email/portal], and requests will be reviewed within [timeframe]. Data will be shared via a secure, restricted-access repository.